CLINICAL TRIAL: NCT02311400
Title: Self-Affirmation, Emotion, and Alcohol Consumption
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999915030; 15-C-N030
Record Dates: First submitted 2014-12-05; First posted 2014-12-08 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2016-09-29

CONDITIONS: Risk Reduction Behavior
Keywords: Emotion; Self-Affirmation; Alcohol Consumption
MeSH Terms: conditions — Risk Reduction Behavior; Alcohol Drinking

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
Background:

- People respond differently to life events and how those events make them feel. They also respond differently to information about the how their actions affect their lives and health. Researchers want to learn more about these differences. In this study, researchers will look at how people respond to an event in their life. Researchers will also look at how people respond to information about how their actions can affect their health.

Objective:

- To see how people respond differently to life events and information about alcohol and breast cancer.

Eligibility:

- Women 18 and older who have never been diagnosed with cancer and who drank 5 or more alcoholic drinks in the past week.

Design:

* This study will take place online.
* Participants will be randomly assigned to 1 of 10 groups.
* Researchers will ask participants to take part in 2 small studies, 1 about Life Events and 1

about Alcohol and Breast Cancer.

* In the Life Events study, participants will write briefly about a time they felt very happy, fearful, angry, or surprised, or they will write about a room in their house. Then they will answer questions about that event. They also will write about a value that is or is not important to them.
* In the Alcohol and Breast Cancer study, participants will read a health message about the link between alcohol and breast cancer. Then they will answer questions about what they read and give their thoughts about alcohol and breast cancer.
* Both studies should take about 30 minutes.

DETAILED DESCRIPTION:
This study aims to examine whether emotional state moderates the effect of selfaffirmation on intentions to engage in proactive behavior following a message about a health threat. Specifically, we propose to examine whether selfaffirmation a process by which individuals reflect on cherished personal values differentially affects the persuasiveness of a message about the link between alcohol and breast cancer depending on whether individuals are in a particular emotional state. Previous evidence suggests that self-affirmation may reduce defensiveness to threatening health information, increasing openness to the message and resulting in increased disease risk perceptions, disease-related worry, and intentions to engage in preventive behavior. However, self-affirmation may be differentially effective depending on the prior emotional state of the individual. Human subjects (women who report having consumed five or more alcoholic beverage in the past week) will be randomly assigned to write about an emotional event (something that made them happy, fearful, angry, or surprised) or to a neutral emotion condition (writing about a room in their house). Then, they will be randomly assigned to selfaffirm (write about why a particular value is important to them) or to be in a control condition (write about why a particular value might be important to someone else). Following the autobiographical emotion task and self-affirmation, subjects will read about the link between alcohol and breast cancer. Finally, they will be asked a series of questions about their intentions to reduce drinking, their perceived risk of breast cancer, and their worry about breast cancer. Drawing on previous research, we hypothesize that self-affirmation will be most effective for those asked to recall a happy or angry experience, and least effective for those asked to recall a fearful or surprising experience.

ELIGIBILITY:
* INCLUSION AND EXCLUSION CRITERIA:

Women who have never been diagnosed with cancer and who drank 5 + alcoholic beverages in the past week will be eligible to participate. All men, and women who report a lower threshold of alcohol consumption, will be excluded.

Children will be excluded from this study.

Participants who have completed prior self-affirmation studies through GfK (e.g., the one conducted under 12-C-N162-B) will also be excluded; these participants will be identified by GfK (based on records of study participation kept for panel members), and will not be invited to participate in the current study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 690 (Actual)
Dates: Start 2014-11-19; Primary Completion 2015-04-01 (Actual); Study Completion 2016-09-29 (Actual)

PRIMARY OUTCOMES:
Alcohol cessation intentions | immediately post-experiment

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca A Ferrer, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- GfK, Menlo Park, California, United States

REFERENCES:
- [Background] Epton T, Harris PR. Self-affirmation promotes health behavior change. Health Psychol. 2008 Nov;27(6):746-52. doi: 10.1037/0278-6133.27.6.746. PMID 19025270
- [Background] Lerner JS, Keltner D. Fear, anger, and risk. J Pers Soc Psychol. 2001 Jul;81(1):146-59. doi: 10.1037//0022-3514.81.1.146. PMID 11474720
- [Background] Harris PR, Napper L. Self-affirmation and the biased processing of threatening health-risk information. Pers Soc Psychol Bull. 2005 Sep;31(9):1250-63. doi: 10.1177/0146167205274694. PMID 16055644